CLINICAL TRIAL: NCT00034957
Title: Study of the Efficacy of an Investigational Drug in Adult Patients With Non Small-Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 196-ONC-0100-005
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Neoplasms
Keywords: Pharmacia
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Drugs, Investigational

INTERVENTIONS:
Drug: Investigational drug

SUMMARY:
The primary goal of the study is to evaluate an investigational drug's effectiveness as a treatment for Non small-cell lung cancer (NSCLC)

ELIGIBILITY:
Other specific inclusion/exclusion criteria may apply. In order to determine eligibility, further examination by the investigator is necessary.

Inclusion Criteria: Eligible patients must be at least 18 years of age with a diagnosis of NSCLC that has gotten worse during or after treatment with platinum-based chemotherapy. Patients must have at least one tumor that can be evaluated by the doctor during the investigational drug treatment. Any side-effects from prior chemotherapy must have subsided, and blood and urine tests must show adequate bone marrow, liver, and kidney function.

Exclusion Criteria: Any of the following will exclude patients from study participation: receipt of more than 1 prior regimen of chemotherapy for NSCLC (repeat of the same chemotherapy at different points in time count as 1 regimen). Irradiation to 25% or more of bone marrow, prior high dose chemotherapy with bone marrow or stem cell support, current participation in other clinical trials, pregnant or breast-feeding women, known HIV-positive or AIDS-related illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Primary Completion 2002-10 (Actual); Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Research Center, Berkeley, California
  - Research Center, Greenbrae, California
  - Research Center, Los Angeles, California
  - Research Center, Rancho Mirage, California
  - Research Center, Chicago, Illinois
  - Research Center, Louisville, Kentucky
  - Research Center, West Boylston, Massachusetts
  - Research Center, Ann Arbor, Michigan
  - Research Center, Lebanon, New Hampshire
  - Research Center, Nashville, Tennessee
  - Research Center, Arlington, Texas
  - Research Center, Dallas, Texas